CLINICAL TRIAL: NCT06532110
Title: The Role of Gut Microbiota in Chronic GI Diseases: A Pilot Study
Brief Title: Gut Microbiota in Chronic GI Diseases
Acronym: ChronicGI
Status: Recruiting | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: HiREB-15311
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Microbiota
Keywords: microbiota; chronic gastrointestinal disorders; colonization; metabolites
MeSH Terms: interventions — Endoscopy; Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic gastrointestinal disorders: A cohort of 260 patients (150 diagnosed with IBD, 40 with IBS, 30 with celiac disease, 10 with MC, 10 with functional diarrhea and 30 non-disease controls) of either sex between 18 and 75 years of age consulting to either the GI Clinical Investigation, the Endoscopy Unit (McMaster University)
  Interventions: Other: Endoscopy/Colonoscopy

INTERVENTIONS:
Other: Endoscopy/Colonoscopy — Esophagogastroduodenoscopy and colonoscopy with video recording and biopsy collection

SUMMARY:
The study involves characterizing the microbiota of patients with IBS, functional diarrhea, IBD, severe motility disorders and celiac disease.

This will be complemented by a translational phase of human-mouse hybrid experiments in which germ-free mice will be colonized with feces from these patients with different GI disease and non-disease controls and we will compare symptoms, microbiota composition and histological changes in the gut and in the brain of the mice.

DETAILED DESCRIPTION:
A complex community of microbes collectively referred to as microbiota, inhabit the human body. The intestinal microbiota is a diverse and dynamic ecosystem, which has developed a mutualistic relationship with its host and plays a crucial role in the development of the host's innate and adaptive immune responses. This ecosystem serves the host by protecting against pathogens, harvesting otherwise inaccessible nutrients, aiding in neutralization of drugs and carcinogens, and affecting the metabolism of lipids. Gut bacteria modulate intestinal motility, barrier function and visceral perception. A better understanding of the role of microbiota in the proposed GI diseases will have profound impact in the characterization of future biomarkers and has also potential treatment implications. As the microbiota may be disturbed in the mentioned GI conditions, a possible treatment approach could be to correct dysbiosis either by the administration of an antibiotic or a preparation of 'beneficial' bacteria (probiotics) according to each bacteria profile.

General Objective The objective of this study is to identify different patterns of intestinal microbiota in patients diagnosed with inflammatory bowel disease, microscopic colitis, functional diarrhea, severe motility disorders, celiac disease and irritable bowel syndrome and to compare it with non-disease controls, by assessing data (questionnaires) and samples (stool, blood and tissue) from single time point (endoscopy/colonoscopy appointment).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD, active celiac disease (aTTG positive + endoscopic view and histological findings compatible), IBS (Rome IV criteria or physician diagnosis) severe motility disorders (severe constipation, severe functional dyspepsia) gluten sensitivity (IBS diarrhea predominant with positive anti gliadin antibodies and negative aTTG), functional diarrhea (Rome IV criteria), anal fissure and/or fistula or non-disease control individual or 1st degree family member of celiac patient.
* Willingness to participate
* Signed Informed Consent

Exclusion Criteria:

* Antibiotics in the last month
* Probiotics in the previous month

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cohort of 260 patients of either sex between 18 and 75 years of age consulting to either the GI Clinical Investigation, the Endoscopy Unit (McMaster University Endoscopy Centre)
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2012-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
To identify different patterns of intestinal microbiota in patients diagnosed with chronic gastrointestinal disorders or controls | October 2013 - October 2026
  To identify different patterns of intestinal microbiota in patients diagnosed with inflammatory bowel disease, microscopic colitis, functional diarrhea, severe motility disorders, celiac disease and irritable bowel syndrome and to compare it with non-disease controls.

SECONDARY OUTCOMES:
To study the effect of microbiota on the immune system | October 2013 - October 2026
  Through colonization of germ free mice with human feces from the different groups of patients and controls.
To compare luminal microbiota composition vs. mucosa-associated microbiota composition in patients diagnosed with IBD, IBS, microscopic colitis, functional diarrhea, severe motility disorders and celiac disease and non-disease controls. | October 2013 - October 2026
  Assessed by stool samples and aspirates, representative to the luminal composition; and the intestinal tissue (biopsies) representative of the mucosa
To assess and compare the metabolic activity of gut bacteria of IBD, IBS, microscopic colitis, severe motility disorders, functional diarrhea and celiac disease patients and non-disease controls | October 2013 - October 2026
  Through assessing different bacteria derived metabolites, such as short-chain fatty acids

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bercik P. The microbiota-gut-brain axis: learning from intestinal bacteria? Gut. 2011 Mar;60(3):288-9. doi: 10.1136/gut.2010.226779. No abstract available. PMID 21296788
- [Result] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Result] Parkes GC, Brostoff J, Whelan K, Sanderson JD. Gastrointestinal microbiota in irritable bowel syndrome: their role in its pathogenesis and treatment. Am J Gastroenterol. 2008 Jun;103(6):1557-67. doi: 10.1111/j.1572-0241.2008.01869.x. Epub 2008 May 29. PMID 18513268
- [Result] Bolino CM, Bercik P. Pathogenic factors involved in the development of irritable bowel syndrome: focus on a microbial role. Infect Dis Clin North Am. 2010 Dec;24(4):961-75, ix. doi: 10.1016/j.idc.2010.07.005. PMID 20937460
- [Result] Collins SM, Denou E, Verdu EF, Bercik P. The putative role of the intestinal microbiota in the irritable bowel syndrome. Dig Liver Dis. 2009 Dec;41(12):850-3. doi: 10.1016/j.dld.2009.07.023. Epub 2009 Sep 8. PMID 19740713
- [Result] Gwee KA, Collins SM, Read NW, Rajnakova A, Deng Y, Graham JC, McKendrick MW, Moochhala SM. Increased rectal mucosal expression of interleukin 1beta in recently acquired post-infectious irritable bowel syndrome. Gut. 2003 Apr;52(4):523-6. doi: 10.1136/gut.52.4.523. PMID 12631663
- [Result] Gwee KA, Leong YL, Graham C, McKendrick MW, Collins SM, Walters SJ, Underwood JE, Read NW. The role of psychological and biological factors in postinfective gut dysfunction. Gut. 1999 Mar;44(3):400-6. doi: 10.1136/gut.44.3.400. PMID 10026328
- [Result] Dunlop SP, Jenkins D, Neal KR, Spiller RC. Relative importance of enterochromaffin cell hyperplasia, anxiety, and depression in postinfectious IBS. Gastroenterology. 2003 Dec;125(6):1651-9. doi: 10.1053/j.gastro.2003.09.028. PMID 14724817
- [Result] Marshall JK, Thabane M, Garg AX, Clark WF, Salvadori M, Collins SM; Walkerton Health Study Investigators. Incidence and epidemiology of irritable bowel syndrome after a large waterborne outbreak of bacterial dysentery. Gastroenterology. 2006 Aug;131(2):445-50; quiz 660. doi: 10.1053/j.gastro.2006.05.053. PMID 16890598
- [Result] Malinen E, Rinttila T, Kajander K, Matto J, Kassinen A, Krogius L, Saarela M, Korpela R, Palva A. Analysis of the fecal microbiota of irritable bowel syndrome patients and healthy controls with real-time PCR. Am J Gastroenterol. 2005 Feb;100(2):373-82. doi: 10.1111/j.1572-0241.2005.40312.x. PMID 15667495
- [Result] Kerckhoffs AP, Samsom M, van der Rest ME, de Vogel J, Knol J, Ben-Amor K, Akkermans LM. Lower Bifidobacteria counts in both duodenal mucosa-associated and fecal microbiota in irritable bowel syndrome patients. World J Gastroenterol. 2009 Jun 21;15(23):2887-92. doi: 10.3748/wjg.15.2887. PMID 19533811
- [Result] Krogius-Kurikka L, Lyra A, Malinen E, Aarnikunnas J, Tuimala J, Paulin L, Makivuokko H, Kajander K, Palva A. Microbial community analysis reveals high level phylogenetic alterations in the overall gastrointestinal microbiota of diarrhoea-predominant irritable bowel syndrome sufferers. BMC Gastroenterol. 2009 Dec 17;9:95. doi: 10.1186/1471-230X-9-95. PMID 20015409
- [Result] Carroll IM, Chang YH, Park J, Sartor RB, Ringel Y. Luminal and mucosal-associated intestinal microbiota in patients with diarrhea-predominant irritable bowel syndrome. Gut Pathog. 2010 Dec 9;2(1):19. doi: 10.1186/1757-4749-2-19. PMID 21143915
- [Result] Tana C, Umesaki Y, Imaoka A, Handa T, Kanazawa M, Fukudo S. Altered profiles of intestinal microbiota and organic acids may be the origin of symptoms in irritable bowel syndrome. Neurogastroenterol Motil. 2010 May;22(5):512-9, e114-5. doi: 10.1111/j.1365-2982.2009.01427.x. Epub 2009 Nov 10. PMID 19903265
- [Result] Nistal E, Caminero A, Vivas S, Ruiz de Morales JM, Saenz de Miera LE, Rodriguez-Aparicio LB, Casqueiro J. Differences in faecal bacteria populations and faecal bacteria metabolism in healthy adults and celiac disease patients. Biochimie. 2012 Aug;94(8):1724-9. doi: 10.1016/j.biochi.2012.03.025. Epub 2012 Apr 20. PMID 22542995
- [Result] Nadal I, Donant E, Ribes-Koninckx C, Calabuig M, Sanz Y. Imbalance in the composition of the duodenal microbiota of children with coeliac disease. J Med Microbiol. 2007 Dec;56(Pt 12):1669-1674. doi: 10.1099/jmm.0.47410-0. PMID 18033837
- [Result] Collado MC, Donat E, Ribes-Koninckx C, Calabuig M, Sanz Y. Imbalances in faecal and duodenal Bifidobacterium species composition in active and non-active coeliac disease. BMC Microbiol. 2008 Dec 22;8:232. doi: 10.1186/1471-2180-8-232. PMID 19102766
- [Result] Collado MC, Donat E, Ribes-Koninckx C, Calabuig M, Sanz Y. Specific duodenal and faecal bacterial groups associated with paediatric coeliac disease. J Clin Pathol. 2009 Mar;62(3):264-9. doi: 10.1136/jcp.2008.061366. Epub 2008 Nov 7. PMID 18996905
- [Result] Sanchez E, Donat E, Ribes-Koninckx C, Calabuig M, Sanz Y. Intestinal Bacteroides species associated with coeliac disease. J Clin Pathol. 2010 Dec;63(12):1105-11. doi: 10.1136/jcp.2010.076950. Epub 2010 Oct 23. PMID 20972239
- [Result] Gillevet P, Sikaroodi M, Keshavarzian A, Mutlu EA. Quantitative assessment of the human gut microbiome using multitag pyrosequencing. Chem Biodivers. 2010 May;7(5):1065-75. doi: 10.1002/cbdv.200900322. PMID 20491064